CLINICAL TRIAL: NCT03194217
Title: Dose Finding Phase IIb Study of Bavisant to Evaluate Its Safety and effiCacy in treAtment of exceSsive Daytime sleePiness (EDS) in PARkinson's Disease (PD).
Brief Title: BEN-2001 in Parkinson Disease Patients With Excessive Daytime Sleepiness
Acronym: CASPAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BenevolentAI Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BB-2001-201b
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Results first posted 2020-11-24 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Excessive Daytime Sleepiness; Parkinson Disease
MeSH Terms: conditions — Disorders of Excessive Somnolence; Parkinson Disease | interventions — bavisant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BEN-2001, 0.5mg (Experimental): Experimental treatment
  Interventions: Drug: BEN-2001
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo
- BEN-2001, 1.0mg (Experimental): Experimental treatment
  Interventions: Drug: BEN-2001
- BEN-2001, 3.0mg (Experimental): Experimental treatment
  Interventions: Drug: BEN-2001

INTERVENTIONS:
Drug: BEN-2001 — Bavisant dihydrochloride monohydrate for oral use
  Other Names: Bavisant
  Arms: BEN-2001, 0.5mg; BEN-2001, 1.0mg; BEN-2001, 3.0mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This phase 2b study is designed as multicentre, multinational, randomized, double blind, parallel group and placebo controlled with three doses of Bavisant (0.5, 1, and 3 mg/d) in subjects with excessive daytime sleepiness with Parkinson's disease.

DETAILED DESCRIPTION:
Phase 2b study will be conducted with the aim of investigating the efficacy and safety of three fixed doses of Bavisant (0.5, 1 and 3 mg/d) compared to placebo for the treatment of excessive daytime sleepiness (EDS) in subjects with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either sex aged 50 to 80 years *Subjects with previous diagnosis of Parkinson's disease (following the UK Parkinson's disease society brain bank clinical diagnostic criteria)*
* Subjects capable of understanding and complying with protocol requirements
* Subjects with medical history of excessive daytime sleepiness

Exclusion Criteria:

* Subjects with excessive daytime sleepiness due to conditions other than Parkinson's disease (including narcolepsy)
* Subjects with clinical evidence of depression with significant psychiatric comorbidities (Hamilton Rating Scale for Depression - HAM-D score greater than or equal to 17; with or without treatment)
* Subjects with evidence of significant fatigue (Fatigue Severity Scale - FSS greater than or equal to 36
* Subjects with known history of abuse of alcohol or other addictive substances in the 6 months prior to inclusion.
* Subjects with known allergies or hypersensitivity to Bavisant or any of its excipients.
* Subjects who are pregnant or lactating.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G Ondo, M.D, Principal Investigator — Methodist Neurological Institute
Locations (1):
- MaxBlue Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | BEN-2001, 0.5mg | BEN-2001, 1.0mg | BEN-2001, 3.0mg
Started | 60 | 60 | 60 | 64
Completed | 60 | 57 | 56 | 60
Not Completed | 0 | 3 | 4 | 4
Not completed — Adverse Event | 0 | 2 | 3 | 3
Not completed — Failure to meet randomisation criteria | 0 | 0 | 0 | 1
Not completed — Other | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BEN-2001, 0.5mg | BEN-2001, 1.0mg | BEN-2001, 3.0mg | Total
Number analyzed (Participants) | 60 | 60 | 60 | 64 | 244
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 21 | 18 | 27 | 84
  >=65 years | 42 | 39 | 42 | 37 | 160
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 17 | 20 | 81
  Male | 39 | 37 | 43 | 44 | 163
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 59 | 57 | 59 | 64 | 239
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 11 | 11 | 47
  Europe | 47 | 48 | 49 | 53 | 197

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Sleepiness Using the Epworth Sleepiness Scale (ESS) at Baseline and Post Dose.
Description: Mean absolute change of Bavisant treatment groups in the Epworth Sleepiness Scale (ESS) from baseline to the end of the 6-week treatment period.
  The ESS score (sum of 8 item scores) ranges from 0 to 24 with higher score corresponding to higher average sleep propensity in daily life (higher daytime sleepiness).
  Eligibility determined based on ESS score of 13 and above.
Time Frame: 6 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | BEN-2001, 0.5mg | BEN-2001, 1.0mg | BEN-2001, 3.0mg
Number analyzed (Participants) | 60 | 60 | 60 | 64
units on a scale | -4.34 (0.5) | -4.64 (0.51) | -3.46 (0.51) | -4.73 (0.5)
Statistical Analysis 1: Comparison: BEN-2001, 0.5mg; Test type: Superiority; p = 0.668, ANCOVA; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-1.68 to 1.08], Standard Error of Mean 0.70
Statistical Analysis 2: Comparison: BEN-2001, 1.0mg; Test type: Superiority; p = 0.213, ANCOVA; Mean Difference (Final Values) = 0.88, 95% CI 2-sided [-0.50 to 2.26], Standard Error of Mean 0.70
Statistical Analysis 3: Comparison: BEN-2001, 3.0mg; Test type: Superiority; p = 0.575, ANCOVA; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-1.76 to 0.98], Standard Error of Mean 0.70

ADVERSE EVENTS:
Time Frame: 70 days
Arm/Group | Placebo | BEN-2001, 0.5mg | BEN-2001, 1.0mg | BEN-2001, 3.0mg
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/60 | 0/64
Serious Adverse Events (participants affected / at risk) | 1/60 | 0/60 | 0/60 | 2/64
Other Adverse Events (participants affected / at risk) | 11/60 | 16/60 | 27/60 | 26/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=60) | BEN-2001, 0.5mg (N=60) | BEN-2001, 1.0mg (N=60) | BEN-2001, 3.0mg (N=64)
cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=60) | BEN-2001, 0.5mg (N=60) | BEN-2001, 1.0mg (N=60) | BEN-2001, 3.0mg (N=64)
Nasopharygitis (Infections and infestations) | 3 | 2 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 2 | 0
Initial Insomnia (Psychiatric disorders) | 2 | 3 | 1 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 3
Middle Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 3
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 2
Head ache (Nervous system disorders) | 0 | 1 | 2 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 2
Cataract Nuclear (Eye disorders) | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 4 | 3
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2
Fatigue (General disorders) | 0 | 1 | 2 | 1
Triglycerous increase (Investigations) | 1 | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT03194217/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT03194217/SAP_001.pdf